CLINICAL TRIAL: NCT06293248
Title: The Effect of Music on Healing in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Music Application in Patients Undergoing Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, SELDA MERT, Principal Investigator, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 77979112
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Nurse's Role; Patient Satisfaction
Keywords: nursing care; recovery; anxiety; pain; vital signs; confor; quality of care
MeSH Terms: conditions — Patient Satisfaction; Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Patients in this group received routine care and no music application was performed.
- Experimental group (Experimental): The patient information form, vital signs registration form, and state-trait anxiety scale were administered to the patients in the music group while they were in the ward before being sent to the CAG laboratory. Afterward, Rast, Acemasiran, and Huseyni music from Classical Turkish Music modes were optionally offered to the patients, and before the CAG procedure (while the patient was waiting for the procedure in the CAG laboratory), the music preferred by the patients was played with headphones for 15-20 minutes in order not to disturb other patients. After CAG, 15 minutes after the patient arrived at the service, he listened to music for 15-20 minutes. Then, the vital signs registration form, state-trait anxiety scale, Perianesthesia Comfort Scale-PCS" and Patient Satisfaction Survey on Nursing Care Quality (PSSNCQ) were applied.
  Interventions: Other: musical application

INTERVENTIONS:
Other: musical application — Rast, Acemasiran, and Huseyni from Classical Turkish Music modes were optionally offered to the patients in the music group, and the patient's preferred music was listened to through headphones for 15-20 minutes before the CAG procedure. Following the interviews, musical genres were arranged as instrumental, without words, at 70 decibels in terms of rhythm and duration, at approximately 60 metronomes per minute, and were played according to the person's preference. Instrumental music was loaded onto the portable MP3 player provided by the researchers.
  Arms: Experimental group

SUMMARY:
This study was planned to examine the effect of music application on recovery in patients undergoing coronary angiography (CAG) and to obtain the opinions of patients and nurses about music.This study was conducted to examine the effect of music application on recovery in patients undergoing CAG and to obtain the opinions of patients and nurses about music.The study was planned as a pre-test, post-test design, single-center, randomized controlled experimental study. The study is planned to be conducted in the CAG unit of a university hospital between July 2023 and December 2023, the study sample will be composed of a total of 210 individuals, 105 in each group (music applied group before and after the procedure = 105, control group = 105) To collect data in the study, the "Patient Information Form", Vital Signs Evaluation Form", "Numerical Rating Scale", State-Trait Anxiety Inventory, "Perianesthesia Comfort Scale" and "Patient Satisfaction Survey on Nursing Care Quality" were used.

DETAILED DESCRIPTION:
In the study, before the patients in the music group (MG) who would undergo planned CAG listened to music, while the patients were in the ward before the procedure; Patient information form, vital signs registration form, numerical rating scale, state-trait anxiety scale were applied, then 15-20 minutes. Music prepared with expert suggestions (Rast, Acemasiran, and Huseyni modes) 15-20 min. was listened to. After the procedure, patients in MG are given 15-20 minutes before being discharged. music was played. Then, the vital signs registration form, Numerical Rating Scale, state-trait anxiety scale, Perianesthesia Comfort Scale, and Patient Satisfaction Survey on Nursing Care Quality were administered for the last time. The specified survey forms were applied to the patients in Control Group before and after the procedure, and they were not allowed to listen to music.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-65,
* being literate,
* having no communication or hearing impairment or neurological-psychiatric disease,
* not taking sedatives before the procedure
* not having undergone PCI before
* being in the waiting room at least 20 minutes before the procedure.

Exclusion Criteria:

* Under the age of 18
* Do not speak Turkish
* Have a hearing problem
* Without a place and time orientation
* Have any psychiatric illness
* Using sedative or analgesic drugs in the last 24 hours
* To be intervened outside the femoral area
* Previous angiography procedure
* Non-volunteer individuals will not be included in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Means of subjective pain scores | before and up to 30 minutes after the coronary angiography
  Numerical Rating Scale was used to measure the pain intensity of the patients. This scale, which aims to determine the pain intensity of patients regarding the procedure area, aims to explain the patient's pain with numbers.It is stated that numerical scales are more widely adopted by patients because they facilitate the definition of pain intensity, facilitate scoring and recording, and are useful in floor and ceiling effect assessment. The form ranging from 0 to 10 was used in the research. In the form, 0 points are considered "no pain", 1-3 points are considered "mild pain", 4-6 points are considered "moderate pain", and 7 and above points are considered "severe pain".
Means of body temperature (0C) | before and up to 30 minutes after the coronary angiography
  It will be measured by the researcher responsible for the application using an infrared thermometer.
Means of systolic blood pressure (mmHg) | before and up to 30 minutes after the coronary angiography
  The measurement on the arm, which is not operated with a digital blood pressure meter, will be made by researcher responsible for the application.
Means of diastolic blood pressure (mmHg) | before and up to 30 minutes after the coronary angiography
  The measurement on the arm, which is not operated with a digital blood pressure meter, will be made by the researcher responsible for the application.
Means of heart rate (/minutes) | before and up to 30 minutes after the coronary angiography
  It will be measured by the researcher responsible for the application with a pulse oximeter in the unprocessed arm.
Means of respiratory rate (/minutes) | before and up to 30 minutes after the coronary angiography
  It will be counted by the researcher responsible for the application by monitoring chest movements for one minute.
Means of oxygen saturation (%) | before and up to 30 minutes after the coronary angiography
  It will be measured by the researcher responsible for the application with a pulse oximeter in the unprocessed arm.
Means of subjective anxiety scores | before and up to 30 minutes after the coronary angiography
  These scales determine state and trait anxiety levels, and include two separate sections consisting of a total of 40 items developed based on the two-factor anxiety concept. The first 20 of these measure the situation-related anxiety level, and the items from 21 to 40 measure the individual's trait anxiety level. It is stated that 20-39 points obtained from the scale are considered as "mild", 40-59 points as "moderate", 60-79 points as "severe anxiety" and 80 points as "panic".
Means of Perianesthesia Comfort Scale Scores | Up to 30 minutes from coronary angiography
  The Perianesthesia Comfort Scale scale which reveals the individual's thoughts, emotions, and self-understanding during the stages of the surgical process, consists of 24 items and the expressions are in Likert type ranging from 1 to 6 points. The highest total score that can be obtained from the scale is 144, and the lowest total score is 24. The average value is determined by dividing the total score obtained by the number of scale items and the result is stated in the 1-6 distribution. The highest total score that can be obtained from the scale is 144, and the lowest total score is 24. The average value is determined by dividing the total score obtained by the number of scale items and the result is stated in the 1-6 distribution. A low score indicates that comfort is bad, and a high score indicates that comfort is good.
Means of Patient Satisfaction Survey on Nursing Care Quality Scores | Up to 30 minutes from coronary angiography
  Patient Satisfaction with Nursing Care Quality Questionnaire (PSNCQQ): This scale which comprises 19 items in total, includes 4 items that evaluate the perception of general satisfaction and are not included in the calculation. A 5-point Likert-type scale is scored between "(5) excellent" and "(1) poor". The PSNCQQ, where two different methods can score, was scored by adding the scores for all items and averaging each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Selda MERT, PhD, Principal Investigator — Kirsehir Ahi Evran University
Locations (1):
- Kocaeli University Hospital, Kocaeli, Umuttepe Campus, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research will be made available through the journal after it is published.